CLINICAL TRIAL: NCT06754839
Title: Clinical Trial Evaluating the Effectiveness and Safety of Percutaneous Left Ventricular Assist Device in Supporting High-risk Percutaneous Coronary Intervention
Brief Title: Clinical Trial of Ventiflow LP Supporting High-risk Percutaneous Coronary Intervention(PCI)
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Suzhou Hearthill Medical Technology Co.,LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XLMD-ZSFZ-QX02
Record Dates: First submitted 2024-12-19; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Coronary Artery Disease; Heart Failure; High-risk PCI
Keywords: High-risk PCI; Percutaneous left ventricular assist device; heart failure
MeSH Terms: conditions — Coronary Artery Disease; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental group(Ventiflow LP) (Experimental)
  Interventions: Device: Percutaneous left ventricular assist device(Ventiflow LP)
- Control Group(VA-ECMO) (Active Comparator)
  Interventions: Device: VA-ECMO

INTERVENTIONS:
Device: Percutaneous left ventricular assist device(Ventiflow LP) — The PCI will be completed with the support of percutaneous left ventricular assist device(Ventiflow LP).
  Arms: Experimental group(Ventiflow LP)
Device: VA-ECMO — The PCI will be completed with the support of Veno-arterial extracorporeal membrane oxygenation (VA-ECMO).
  Arms: Control Group(VA-ECMO)

SUMMARY:
The purpose of this prospective, multicenter, randomized controlled clinical trial is to evaluate the effectiveness of the transcatheter left ventricular assist system (Ventiflow LP) in providing circulatory support to patients during high-risk PCI procedures compared to veno-arterial extracorporeal membrane oxygenation (VA-ECMO).The participants will be randomly assigned to the experimental group or the control group after enrollment, and will undergo percutaneous coronary intervention(PCI) with support from Ventiflow LP or VA-ECMO respectively. All participants need to undergo a 3-month follow-up after operative.

ELIGIBILITY:
Inclusion Criteria:

1. 18 Years to 90 Years
2. The cardiac team determined that the subject needs coronary artery revascularization, but there is a higher risk of CABG, or the subject refuses to accept CABG. After comprehensive evaluation by the cardiac team, it was determined that the subjects could benefit from PCI
3. The subject is diagnosed with acute or chronic coronary syndrome, and

   1. LVEF≤ 35% or
   2. LVEF ≤ 40% and NYHA Classification is III or IV
4. Informed consent
5. The participant meets all the above clinical inclusion criteria and must comply with at least one of the following imaging criteria.

1. At least two coronary artery CTOs (diameter of occluded artery ≥ 2.5mm) 2. Unprotected left main coronary artery disease, and meeting one or more complex operating standards 3. Three-vessel disease and meeting two or more complex operating standards

Complex operations are defined as:

1. Bifurcation lesions require treatment of dual branches (including stents and PTCA)
2. Calcification lesions require complex operation or instrument assistance (Excimer laser coronary atherectomy, intravascular lithotripsy, or rotational atherectomy)
3. Severe distortion requires complex operations
4. The target lesion is CTO (diameter of occluded artery ≥ 2.5mm and J-CTO score ≥ 2 )

Exclusion Criteria:

1. Acute ST-elevation myocardial infarction within 7 days or receiving thrombolytic therapy;
2. Cardiopulmonary resuscitation within 24 hours;
3. Patients who have had cardiogenic shock (systolic blood pressure < 90 mmHg for more than 30 minutes or need catecholamines to maintain systolic blood pressure above 90 mmHg) or hemodynamic instability within 7 days before surgery;
4. Atrial or ventricular septal defect (including post-infarct VSD), left ventricular wall thrombus; left ventricular rupture, cardiac tamponade, or concomitant cardiopulmonary failure;
5. Presence of aortic stenosis/calcification (aortic orifice area ≤ 0.6cm2), documented moderate to severe aortic regurgitation (echocardiographic assessment grade ≥2+); have an artificial aortic valve;
6. Severe pulmonary hypertension, right heart failure or severe tricuspid regurgitation;
7. Prior or current use of a persistent left ventricular assist device (LVAD), or use of IABP, extracorporeal membrane oxygenation (ECMO), or percutaneous ventricular assist device (such as Impella or Tandem Heart) within 7 days prior to surgery;
8. History of stroke or transient ischemic attack within 1 month before surgery;
9. Patients with renal failure (creatinine ≥3 times ULN) and may require dialysis treatment;
10. Subject has abnormal liver function (elevated aspartate aminotransferase (AST), alanine aminotransferase (ALT) and bilirubin levels ≥3 times ULN);
11. Moderate and severe anemia (hemoglobin <90g/L); Subject has abnormalities in coagulation parameters that cannot be corrected (defined as platelet count ≤ 75×109/L or INR ≥2.0 or fibrinogen ≤1.50g/l); or inability to be treated with antiplatelet agents and anticoagulants;
12. Active visceral hemorrhage within 1 month;
13. History of allergy to heparin, contrast media, etc.;
14. Aortic abnormalities that preclude surgery, including aneurysms, extreme curvature, or calcification; or known severe arterial disease that precludes the trial, such as aortic dissection, Marfan syndrome, etc.;
15. Severe peripheral arterial obstructive disease (stent, tortuosity, stenosis, dissection, etc.) that prevents study device placement;
16. Infection at the site of the planned surgical puncture site or suspected active systemic infection with fever or need for antibiotic therapy;
17. Pregnant women and lactating women;
18. The subject has participated in other medical device clinical trials/drug clinical trials during the same period;
19. ECMO cannot be implanted or there are contraindications to its application and any other conditions that the investigator considers inappropriate to participate in this trial.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2024-12 (Estimated); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of major adverse events within 30 days post-operation. | 30 days post-operation
  Major adverse events are defined as death, stroke, myocardial infarction, revascularization, rehospitalization due to cardiovascular reasons, bleeding types 3, 4, 5 defined by mechanical circulatory support academic research consortium (MCS-ARC) , acute kidney injury, serious device-related adverse events, cardiopulmonary resuscitation.

SECONDARY OUTCOMES:
Incidence of major adverse events within 90 days post-operation. | 90 days post-operation
Incidence of major adverse cardiovascular and cerebrovascular events (MACCE) at 30 days post-operation. | 30 days post-operation
  MACCE is defined as all-cause mortality, myocardial infarction, stroke, and any subsequent revascularization procedures .
Incidence of major adverse cardiovascular and cerebrovascular events (MACCE) at 90 days post-operation. | 90 days post-operation
  MACCE is defined as all-cause mortality, myocardial infarction, stroke, and any subsequent revascularization procedures .
Success rate of hemodynamic support during device use | 90 days post-operation
  definition of successful hemodynamic support: successful delivery and initiation of the device, no hemodynamic deregulation occurs during the device support period (haemodynamic derangement refers to: mean arterial pressure(MAP ) less than 60 mmHg for more than 10 minutes and requires additional vasoactive drug therapy)
The success rate of percutaneous coronary intervention(PCI) | 90 days post-operation
  The success rate of PCI is defined as: residual stenosis < 30% after stent implantation or < 50% after balloon angioplasty, or thrombolysis in myocardial infarction(TIMI) flow grade 3.
Complete revascularization rate | Immediately after the intervention
  Complete revascularization rate is defined as: residual SYNTAX score ≤8
Change in creatinine clearance | Baseline to 48 hours postoperation and 30 days post-operation
The change in left ventricular ejection fraction (LVEF) compared to baseline | Baseline to 30 days post-operation and 90 days post-operation
The change in New York heart association(NYHA) classification compared to baseline | 30 days post-operation, 90 days post-operation
  The NYHA classification of heart function consists of four levels, ranging from I to IV, with heart function progressively deteriorating.
Length of hospital stay within 30 days post-operation | 30 days post-operation
Length of intensive care unit(ICU)/(coronary care unit)CCU stay within 30 days post-operation | 30 days post-operation
Success rate of device operation | 30 days post-operation
  The system has delivered to the designated position and completed the pump start-up without any device failure.
Usage time of research device | 30 days post-operation
  The time from the start to the stop of the research device.
Device performance evaluation | Intraoperation
  The operator scores the device after use, with 5 being the best and 1 being the worst.
The failure rate of the device | Intraoperation
  The failure rate of the device is defined as any component of the research equipment (Ventiflow LP or ECMO) system that is unable to operate according to its designed performance specifications .
Incidence of serious adverse events | 90 days post-operation
  Incidence of serious adverse events: Serious adverse events refer to those that occur during the clinical trial process and result in death or a significant deterioration in health status, including fatal diseases or injuries, permanent impairment of bodily structure or function, and events that require medical or surgical intervention to prevent permanent impairment of bodily structure or function, among others.
The incidence of serious adverse events | 90 days post-operation
  The incidence of serious adverse events related to medical devices: including but not limited to cardiac structural damage, severe limb ischemia (pallor, pulselessness, and necrosis), infections, damage to the aorta and aortic valve, hemolysis, complications requiring surgical intervention, and events leading to subject mortality, permanent or severe disability, significantly prolonged hospitalization, or the need for surgical intervention .

CONTACTS AND LOCATIONS:
Overall Officials: Yujie Zhou, MD, Study Chair — Beijing Anzhen Hospital; Yong He, MD, Study Chair — West China Hospital

IPD SHARING:
Plan to Share IPD: No